CLINICAL TRIAL: NCT00735735
Title: Study of the Measurement of Substance P in the Saliva of Patients With Low Back Pain
Brief Title: Measurement of Substance P in Saliva of Low Back Pain Patients
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: Kovacs Foundation (Other)
Responsible Party: Principal Investigator, Francisco M. Kovacs, Director of Scientific Department, Kovacs Foundation, Kovacs Foundation
Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: FK 26
Record Dates: First submitted 2008-08-14; First posted 2008-08-15 (Estimated); Last update posted 2019-08-28 (Actual); Status verified 2019-08

CONDITIONS: Low Back Pain
Keywords: low back pain; chronic; Substance P
MeSH Terms: conditions — Low Back Pain; Bronchiolitis Obliterans Syndrome

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Other: The taking of a saliva sample from each subject. — After taking the sample, the saliva will be transferred via a pipette to a clean tube which will be labeled with the subject's name, the date and the hour. Once a month the tubes will be sent to the collaborating laboratory for analysis.

SUMMARY:
The purpose of this study is to compare the levels of Substance P in saliva, in patients with severe chronic low back pain and in subjects without it. In addition, to explore a possible cutoff point, in order to define normal and pathological levels of Substance P in saliva. The ultimate objective would be to design a measurement method for use in routine clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Patients referred to the Kovacs Back Pain Unit in Palma de Mallorca for chronic low back pain
* A pain level of 6 or greater on the PI-NRS scale (0=no pain, 10= worst pain possible)
* Seen at the Unit between 9 and 13 hours (due to the circadian rhythm of Substance P in saliva and to avoid great variability in the results)

For healthy subjects:

* Volunteers with no pain (anywhere)
* That in the past year have had no more than 40 days with pain, and no episode of more than 7 days of continuous pain.

Exclusion Criteria:

* Subjects with pain that is additional to or different from chronic low back pain

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2009-02; Primary Completion 2012-01 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Levels of Substance P in the saliva | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Francisco M Kovacs, MD, PhD, Study Director — Kovacs Foundation, Palma de Mallorca, 07012, Spain; Mario Gestoso, MD, Principal Investigator — Kovacs Foundation,Palma de Mallorca, Spain
Locations (1):
- Kovacs Foundation, Palma de Mallorca, Balearic Islands, Spain

REFERENCES:
- [Background] LeVasseur SA, Gibson SJ, Helme RD. The measurement of capsaicin-sensitive sensory nerve fiber function in elderly patients with pain. Pain. 1990 Apr;41(1):19-25. doi: 10.1016/0304-3959(90)91104-Q. PMID 2162020
- [Background] Morton CR, Hutchison WD. Release of sensory neuropeptides in the spinal cord: studies with calcitonin gene-related peptide and galanin. Neuroscience. 1989;31(3):807-15. doi: 10.1016/0306-4522(89)90443-0. PMID 2480554
- [Background] Kowalski ML, Sliwinska-Kowalska M, Kaliner MA. Neurogenic inflammation, vascular permeability, and mast cells. II. Additional evidence indicating that mast cells are not involved in neurogenic inflammation. J Immunol. 1990 Aug 15;145(4):1214-21. PMID 1696295
- [Background] Thomas KL, Andrews PV, Khalil Z, Helme RD. Substance P induced hydrolysis of inositol phospholipids in rat skin in an in vivo model of inflammation. Neuropeptides. 1989 Apr;13(3):191-6. doi: 10.1016/0143-4179(89)90091-7. PMID 2469033